CLINICAL TRIAL: NCT04656808
Title: Guilt Feelings, Dysfunctional Thoughts, Cultural Values and Mental and Physical Health of Dementia Family Caregivers: Longitudinal, Intervention and Experimental Analysis
Brief Title: Guilt Focused Psychological Intervention
Acronym: LONG-CARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Andrés Losada Baltar, Full Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSI2015-65152-C2-1-R
Record Dates: First submitted 2020-11-29; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Guilt; Depressive Symptoms; Anxious Symptoms; Stress, Physiological
Keywords: Caregivers; Dementia; Depression; Anxiety; Stress; Guilt; Psychotherapy
MeSH Terms: conditions — Depression; Dementia; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two treatment conditions
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and assessors are blinded to the study research objectives and aims and to the available and obtained treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guilt focused intervention (Experimental): Following literature on factors associated with guilt experiences in caregivers (Gonyea et al., 2008; Gallego-Alberto et al., 2019; Losada et al., 2014; Prunty & Foli, 2019; Romero-Moreno et al., 2014; Spillers et al., 2008) and previous intervention studies testing an Acceptance and Commitment Therapy intervention for dementia family caregivers (Losada et al., 2015; Márquez-González et al., 2020), a guilt focused intervention was specifically designed for caregivers who experienced high levels of guilt and emotional distress. The program is based on CBT (Márquez-González et al., 2007) and Acceptance and Commitment Therapy (ACT) approaches (Losada et al., 2005; Márquez-González et al., 2010), combined with techniques of Compassion-Focused Therapy (CFT; Gilbert, 2009), which were adapted to work with guilt experienced by family dementia caregivers.
  Interventions: Behavioral: Guilt Focused Intervention
- Cognitive behavioral therapy (Active Comparator): Following the cognitive behavioral model adapted to caregiving (Losada et al., 2006) and considering other previous CBT intervention studies with dementia caregivers (Gallagher-Thompson et al., 2003), a CBT intervention developed and tested for dementia family caregivers (Márquez-González et al., 2007) was used for this study. Specifically, this intervention consists of different components that are described in more detail in Losada et al. (2011) and Márquez-González et al. (2007): a) a cognitive restructuring module aimed at modifying caregivers' dysfunctional thoughts about caregiving into other, more appropriate thoughts which promote the use of more adaptive coping strategies for caregivers; b) increasing pleasant activities or behavioral activation; c) asking for help skills; and d) relaxation techniques for reducing physiological activation.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Guilt Focused Intervention — Psychotherapy, group intervention
  Arms: Guilt focused intervention
Behavioral: Cognitive behavioral therapy — Psychotherapy, group intervention
  Arms: Cognitive behavioral therapy

SUMMARY:
Participants in the intervention study will be 120 caregivers with guilt feelings linked with care and high levels of emotional distress (anxiety and/or depression), randomly allocated to the intervention conditions: intervention group and cognitive-behavioral comparison group. The intervention will be provided in a group setting and will consist in 8 sessions plus 3 booster sessions. The effect of the intervention on guilt feelings, depressive and anxious symptomatology, and biomarkers of cardiovascular risk will be assessed after the intervention and at follow-ups at 6 months.

DETAILED DESCRIPTION:
1. Contact with collaborator centers. Centers with previous collaboration with the research team will provide contact data of potential participants. In addition, information of the project will be made available through posters, news, and internet (e.g., social networks).
2. Previous to the assessment each participant will be randomly allocated to the intervention conditions (guilt focused intervention (GFI) and cognitive behavioral therapy (CBT)) following the CONSORT recommendations. Randomization will be made through random numbers using computerized procedures.
3. Once contacted, caregivers will be requested to sign an informed consent and, if the inclusion criteria are met, the interview will take place. Interviews will be conducted by trained psychologists blinded to the project aims and hypothesis.
4. The interviews will consist in questions and questionnaires specifically selected for the project.
5. The intervention conditions have been developed following previous studies by the team or recognized researchers, or following previous research studies in the topic of caregiving stress or related topics (e.g. psychotherapeutic strategies for reducing distress).
6. The interventions will take place in group format (maximum 8 participants per group). Each intervention will consist in 8 weekly sessions plus 3 booster sessions in a 5 month period.
7. Participants will be assessed again after the intervention (2 months) and at the follow-up (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Identifying themselves as the main caregiver of the relative with dementia
* Dedicating at least one daily hour to caregiving tasks
* Having cared for at least three consecutive months
* Not having participated in a psychotherapeutic intervention in the last year
* Showing scores equal or higher than 16 on the Center for Epidemiological Studies-Depression Scale (CES-D; Radloff, 1977) and/or 13 on the Tension-Anxiety subscale from the Profile of Mood States scale (POMS; McNair et al., 1971)
* Showing a score of at least 16 in the Caregiver Guilt Questionnaire (Losada et al., 2010).

Exclusion Criteria:

* Those different to the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Guilt symptoms | Pre-intervention, post-intervention (two months after the intervention) and follow-up (6 months after the intervention)
  Caregivers' feelings of guilt are measured using the Caregiver Guilt Questionnaire (Losada, A., Márquez-González, M., Peñacoba, C., & Romero-Moreno, R., 2010)
Depressive symptoms | Pre-intervention, post-intervention (two months after the intervention) and follow-up (6 months after the intervention)
  The Center for Epidemiological Studies-Depression Scale (CES-D; Radloff, 1977) is used
Anxiety symptoms | Pre-intervention, post-intervention (two months after the intervention) and follow-up (6 months after the intervention)
  Caregivers' symptoms of anxiety are measured through the Tension-Anxiety subscale from the Profile of Mood States (POMS; McNair, Lorr, & Droppleman, 1971)

SECONDARY OUTCOMES:
Caregiving stressors | Pre-intervention, post-intervention (two months after the intervention) and follow-up (6 months after the intervention)
  Care-recipients' behavioral and psychological symptoms were measured with the disruptive behaviors subscale of the Revised Memory and Behavior Problems Checklist (RMBPC; Teri, 1992)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Alcorcón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under request to the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once the study is published
Access Criteria: Upon request to the Principal Investigator